CLINICAL TRIAL: NCT04176237
Title: A Novel Intervention to Improve Sun Exposure Awareness and Behavior in Children
Brief Title: School-based Randomized Trial of SunSmart Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Myles Cockburn, Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HS-11-00677
Record Dates: First submitted 2019-11-21; First posted 2019-11-25 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Skin Neoplasm
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Intervention Model Description: Schools are randomized to receive one of three conditions: (1) Intervention (the expanded SunSmart program); (2) Control (regular SunSmart program); (3) Observation only. Schools in groups (2) and (3) receive the expanded SunSmart program at the conclusion of their participation in data collection.
Who Masked: Participant
Masking Description: Children in schools do not know which arm they are in. Schools and Investigators do know which arm a school is in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention (Experimental): Schools receive 3 one hour lessons on sun safety, followed by a 1 hour UV dosimtery laboratory session.
  Interventions: Other: UV Dosimetry Laboratory
- Control (No Intervention): Schools receive 3 one hour lessons on sun safety.
- Observation (No Intervention): Schools do not receive any lessons.

INTERVENTIONS:
Other: UV Dosimetry Laboratory — The UV Dosimetry Laboratory is a one hour lesson that incorporates science and health education - kids hypothesize what UV levels will be around the school yard, go and measure UV, review their results, and then come up with a SunSmart plan for playing in the school yard.
  Arms: Intervention

SUMMARY:
The objective of this study is to test a novel classroom-based intervention to motivate youth to limit their sun exposure. The intervention will make the process of learning about sun exposure more person-centered using individual dosimetry readings and feedback that will lead to individual plans for reducing sun exposure.

DETAILED DESCRIPTION:
Childhood sun exposure not only increases melanoma risk, but may establish lifetime patterns of exposure and protection. Individuals receive a substantial proportion of lifetime exposure to ultraviolet radiation (UVR) during childhood, and severe sunburns before age 20 may increase lifetime risk of developing melanoma. The objective of this study is to test a novel classroom-based intervention to motivate youth to limit their sun exposure. The intervention will make the process of learning about sun exposure more person-centered using individual dosimetry readings and feedback that will lead to individual plans for reducing sun exposure. Building on the previously existing SunSmart program the investigators have been conducting in 20 local Los Angeles schools in partnership with USC's Joint Education Project (JEP), this study will implement a Randomized Controlled Trial among 5th-6th graders (aged 10-14), comparing this new education-feedback approach to the existing SunSmart education-only program, testing knowledge, attitudes and behavior before and after the intervention. In a subset of students, the investigators will collect real time UV exposure data using personal dosimetry as a Gold Standard measure of change in UV exposure behaviors. The study design randomizes at least 18 schools to 9 intervention or 9 non-intervention (control) schools, and students within each school all have pre- and post-tests. The investigators will also select classrooms from each school across conditions to have students wear dosimeters pre- and post- Intervention/Control. Using a hierarchical cluster analysis with the school unit taken as random and students as repeated measures within school, the investigators will test the primary hypothesis that improvements in sun exposure behaviors are significantly higher than baseline at post-test in the Intervention than Control group, and that this may even occur without significant differences in sun exposure knowledge and attitudes between the two groups. The investigators will additionally test the hypothesis that total UV exposures obtained from UV dosimetry are significantly lower than baseline in the Intervention than control group after Intervention.

ELIGIBILITY:
Inclusion Criteria:

* Child in classrooms from selected schools in the Los Angeles metropolitan area.

Exclusion Criteria:

* All children will participate in the educational activities, unless they opt out of pre- and post-test questionnaires or are absent from school for any of the education sessions.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3750 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2017-01-10 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Change in sun exposure behavior | One week after completion of education activities
  Self reported change in sun exposure behavior using 4 questions in a self-completed questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Myles G Cockburn, PhD, Principal Investigator — University of Southern California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Miller KA, Huh J, Piombo SE, Richardson JL, Harris SC, Peng DH, Cockburn MG. Sun protection changes among diverse elementary schoolchildren participating in a sun safety intervention: A latent transition analysis of a randomized controlled trial. Prev Med. 2021 Aug;149:106601. doi: 10.1016/j.ypmed.2021.106601. Epub 2021 May 7. PMID 33971211